CLINICAL TRIAL: NCT05240157
Title: Incidence and Outcome of Sepsis in Respiratory Intensive Care Unit
Brief Title: Sepsis in Respiratory Intensive Care Unit
Acronym: SepsisinRICU
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ashraf A Elmaraghy, Associate Professor of Pulmonology, Ain Shams University
Other Study IDs: FMASU MS282/2019
Record Dates: First submitted 2022-01-25; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Aspiration; Mucus in Respiratory Tract
Keywords: Sepsis, SOFA score, Respiratory ICU
MeSH Terms: conditions — Sepsis | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Corticosteroid Derivatives — observational
  Other Names: antibiotics

SUMMARY:
Sepsis is the most common cause of death in non coronary intensive care units (ICUs). In the past 2 decades, the world has witnessed significant increase in the occurrence rate of sepsis (1).

In the ICU, sepsis maybe community acquired (already present on admission) or hospital acquired (obtained during ICU stay).

This study will add adequate data about incidence and outcome of sepsis in Respiratory Intensive Care Unit.

DETAILED DESCRIPTION:
Objective: assessing the incidence and outcome of sepsis in Respiratory Intensive Care Unit, providing a crucially important data to increase awareness of the impact of sepsis and highlighting the need for continued research into potential preventive and therapeutic interventions.

Patients and Methods:

This prospective observational cohort study was conducted upon patients admitted at Respiratory Intensive Care Unit (RICU) of Abbassia Chest Hospital, Cairo, Egypt, either with sepsis or acquired sepsis in the RICU; from 1st of May 2019 to 30th of November 2019.

o Inclusion Criteria: Patients ≥ 18 years old with sepsis or septic shock either on admission or acquired at RICU and all episodes of sepsis for the same patient were counted.

o Exclusion Criteria: Patients with length of stay (LOS) at RICU less than 24 hours, patients readmitted at RICU during the same hospitalization, patients admitted at RICU post cardiac arrest, or patients with malignancies.

Data collection and recording:

On admission, the following was done and recorded for all participants:

1. Detailed medical history; including history of previous ICU admission or mechanical ventilation, last antibiotic intake, infected intra venous (IV) or central venous (CV) lines, associated comorbidities and reason of ICU admission.
2. Full general and local chest clinical examination.
3. Need for vasoactive therapy, fluid balance and need for renal replacement therapy.
4. Laboratory investigations:

   * Complete blood picture (CBC).
   * Arterial blood gases analysis (ABGs) on a daily basis.
   * Serum Sodium (Na) and Potassium (K).
   * Liver and Kidney function tests.
   * Serum lactate (repeated when needed to fulfill criteria for diagnosis of septic shock).
5. Radiological investigations;

   * Chest X ray (CXR).
   * Computed Tomography chest, or brain (when appropriate).
6. Microbiological samples culture and sensitivity (when appropriate): Sputum, urine, pleural fluid, or from infected IV line according to the suspected site. Type of infection (community or hospital acquired), infection site: (lungs, urinary tract, abdomen, surgical wound), pathogenic organisms (gram positive, gram negative, atypical bacteria and fungi) were recorded.
7. Scores:

   1. Quick Sequential Organ Failure Assessment (qSOFA) score was recorded at emergency room. (3)
   2. Sequential Organ Failure Assessment (SOFA) score was recorded upon RICU admission and on 3rd and 7th day of ICU stay. (4)
   3. Acute Physiology and Chronic Health Evaluation (APACHE II) score was recorded within 24 hours from patient RICU admission. (3,5)
8. Recording of following points:

   * Number of patients who were on mechanical ventilation, length of RICU stay, presence of comorbidities, survived patients and dead ones, as regards causes of death and risk factors.
   * Complications e.g., acute respiratory distress syndrome (ARDS), acute kidney injury (AKI), septic shock.

Measured Outcomes:

* Primary: Incidence of sepsis, mortality from sepsis.
* Secondary: RICU length of stay due to sepsis, complications from sepsis, mechanical ventilation due to sepsis, need for vasoactive agents.
* Total RICU mortality was also recorded.

Management:

All patients were subjected to the following management protocol regarding the recent Surviving Sepsis Campaign Bundle Update (6):

1. Measuring lactate level with serial measurement if it was more than 2 mmol/L.
2. Blood culture prior to antibiotic administration.
3. For patients with sepsis, early empiric broad-spectrum antibiotic therapy initiated antimicrobial coverage included either an extended spectrum beta lactam, a third or fourth generation cephalosporin, or a carbapenem. Additional consideration was paid to methicillin resistant Staphylococcus aureus (MRSA) risk factors and if present, empiric vancomycin administration was advised. Widespread use of combination therapy, the use of multiple antibiotics with different pharmacodynamic profiles and mechanisms of action reported a synergistic effect with the addition of an aminoglycoside to a beta- lactam Combination therapy has been shown to improve survival. Patients with a high risk of mortality such as septic shock received a combination therapy with at least two different classes of antibiotics depending on type of organism, source of infection, choice of antibiotics kept in mind the most organisms isolated from septic patients.
4. Early fluid resuscitation using 30 mL/Kg crystalloid fluid was given for cases of hypotension or when lactate level > 4mmol/L.
5. Perfusion assessment using CVP and central venues oxygen saturation.
6. Vasopressor use (norepinephrine was given) for persistent hypotension to maintain MAP ≥ 65 mmHg.
7. Adjunctive therapy with steroids (200 mg IV hydrocortisone/day) was given in patients with sepsis who remain hemodynamically unstable despite adequate fluid resuscitation and vasopressor therapy.
8. Glycemic control was done when patient's blood glucose level exceeded 180 mg/dL by administrating insulin.

Study tools and definitions:

The sequential organ failure assessment (SOFA) score was used to demonstrate organ dysfunction (4). Sepsis was defined as having SOFA score of 2 or more plus evidence of infection. Septic shock was defined when persistent hypotension required the use of vasopressors to maintain a MAP ≥ 65 mmHg, and a serum lactate > 2 mmol/L that persisted despite adequate fluid resuscitation. (4) Infection was suspected and confirmed from history, examination, laboratory, radiological and microbiological investigations. ICU acquired infection was defined as infection identified at least 48 hours after ICU admission, while non-ICU acquired infection was defined as infection presented on admission or within the first 48 hours after ICU admission. (7) ARDS was defined according to Berlin definition (8). Acute kidney injury was defined as an abrupt (within hours) decrease in kidney function based on an acute decrease of glomerular filtration rate, as reflected by an acute rise in serum creatinine levels and/or a decline in urine output over a given time interval. (9)

Statistical Analysis:

Data were collected, revised, coded and entered to the Statistical Package for Social Science (IBM SPSS) version 23. The quantitative data were presented as mean, standard deviation, frequency (number of cases and percentage) and ranges when their distribution found parametric and median with interquartile range when their distribution found non-parametric. Qualitative variables were presented as number and percentages. Comparison of numerical variables between the study groups was done using student t- test and paired t-test. The comparison of categorical data was done by using Chi-square test. The level of significance was taken at p value ≤ 0.05 as follows: p > 0.05: non-significant, p < 0.05: significant and p < 0.01: highly significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old with sepsis or septic shock either on admission or acquired at RICU and all episodes of sepsis for the same patient were counted.

Exclusion Criteria:

* Patients with length of stay (LOS) at RICU less than 24 hours, patients readmitted at RICU during the same hospitalization, patients admitted at RICU post cardiac arrest, or patients with malignancies

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted at Respiratory Intensive Care Unit (RICU) of Abbassia Chest Hospital, Cairo, Egypt, either with sepsis or acquired sepsis in the RICU
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of sepsis | 6 months
  Outcome of sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf M Madkour, Prosessor, Study Chair — Ain Shams University
Locations (1):
- Abbassia Chest Hospital, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: No
No sharing of patients data